CLINICAL TRIAL: NCT07396974
Title: Increasing Treatment Access in Trauma Exposed Children: Developing an Adapted Step One Intervention (RCT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Child Mental Health Care Consortium (Unknown); Baylor College of Medicine (Other); University of South Florida (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Leslie Taylor, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-25-0929 (RCT)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Trauma; Posttraumatic Stress Disorder
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Stepped Care Cognitive Behavioral Therapy for Children after Trauma (pSC-CBT-CT) (Experimental): The SC-CBT-CT intervention in this study is a data driven, stakeholder-informed revision of SC-CBT-CT that incorporates Latino specific values and beliefs, that is, personalized SC-CBT-CT (pSC-CBT-CT). The intervention consists of two steps utilizing Cognitive Behavioral Therapy (CBT). Step one (Stepping Together for Children after Trauma, SC-CT) involves a caregiver-led, therapist-assisted first step with narrative, imaginal, and exposure therapy, and step two consists of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT), which utilizes gradual exposure. SC-CT includes three therapist-led caregiver-child meetings over 6-9 weeks, with brief weekly phone support (10-15 minutes) from the therapist to caregiver. During 11 home-based, caregiver-led meetings, the child and caregiver work together on therapeutic tasks (i.e., exposure tasks, a trauma narrative, and in-vivo exposure reminders) guided by an empirically supported activity book.
  Interventions: Behavioral: Personalized Stepped Care Cognitive Behavioral Therapy for Children after Trauma (pSC-CBT-CT)
- Treatment as Usual (TAU) (Active Comparator): Participants in the TAU condition will be given a list of community resources offering child mental health services for trauma survivors. TAU will likely be Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) or another trauma-informed psychotherapy, which may include similar components.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Personalized Stepped Care Cognitive Behavioral Therapy for Children after Trauma (pSC-CBT-CT) — The SC-CBT-CT intervention in this study is a data driven, stakeholder-informed revision of SC-CBT-CT that incorporates Latino specific values and beliefs, that is, personalized SC-CBT-CT (pSC-CBT-CT). The intervention consists of two steps utilizing Cognitive Behavioral Therapy (CBT). Step one (Stepping Together for Children after Trauma, SC-CT) involves a caregiver-led, therapist-assisted first step with narrative, imaginal, and exposure therapy, and step two consists of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT), which utilizes gradual exposure. SC-CT includes three therapist-led caregiver-child meetings over 6-9 weeks, with brief weekly phone support (10-15 minutes) from the therapist to caregiver. During 11 home-based, caregiver-led meetings, the child and caregiver work together on therapeutic tasks (i.e., exposure tasks, a trauma narrative, and in-vivo exposure reminders) guided by an empirically supported activity book.
  Arms: Personalized Stepped Care Cognitive Behavioral Therapy for Children after Trauma (pSC-CBT-CT)
Behavioral: Treatment as Usual (TAU) — Participants in the TAU condition will be given a list of community resources offering child mental health services for trauma survivors. TAU will likely be Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) or another trauma-informed psychotherapy, which may include similar components.
  Arms: Treatment as Usual (TAU)

SUMMARY:
One of the most common and widely disseminated trauma treatments is Trauma Focused Cognitive Behavioral Therapy (TF-CBT). TF-CBT is a therapist-led, structured and sequential intervention, with treatment organized around P.R.A.C.T.I.C.E. (Psychoeducation, Parent training, Relaxation, Affective Regulation, Cognitive Coping, Trauma Narrative, In-Vivo Exposure, Cognitive Reprocessing, and Enhancing Safety) components. Stepped Care Cognitive Behavioral Therapy for Children after Trauma (SC-CBT-CT) is an alternative delivery system that incorporates the best available evidence on the treatment of childhood Post-traumatic Stress Disorder (PTSD) within a stepped care model and utilizes task-shifting with caregiver involvement, which engages caregivers in actively helping their children. Stepped care approaches are characterized by a personalized approach to care in which a lower intensity (i.e., fewer number of sessions) intervention is initially provided before the child is reevaluated or ''stepped up'' for additional care should symptoms persist. The goal of this study is to assess a personalized modification of SC-CBT-CT for Latino families (pSC-CBT-CT). The hypothesis is that personalizing SC-CBT-CT will improve outcomes for Latino children.

ELIGIBILITY:
Inclusion Criteria:

* parent and child agree that the target event/index trauma occurred;
* report of at least five symptoms of PTSD (1 from re-experiencing category or 1 from avoidance);
* suicidal ideation does not exclude as long as there is no active plan/intent. Safety planning implemented and continued assessment for plan/intent;
* children ages 7-12 and a legal guardian willing to participate;
* can be fluent in English or Spanish;
* at least 4 weeks since child's exposure to one or more potentially traumatic events;
* trauma exposure occurred after child was 36 months old.

Exclusion Criteria:

* Children with pervasive developmental disorders or Autism;
* legal guardian or child with active psychosis;
* any condition that may limit the legal guardian ability to understand CBT and the child's ability to follow instructions;
* children who have unsupervised visitation with their perpetrator;
* perpetrator (person that harmed child) is living in the home;
* active substance use disorder;
* child is currently receiving trauma-focused therapy;
* legal guardian is actively suicidal will be excluded from participation;
* children who have not been stable on psychotropic medication for 4 or more weeks, and/or for benzodiazepines/stimulants not stable for 2 or more weeks will not be eligible for the trial.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Stress Severity and Impairment as Assessed by the UCLA PTSD Reaction Index (RI) for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (UCLA-RI-5) - Child Reported | baseline, week 7, week 15
  Total score ranges from 0 to 73, with a higher score indicating worse symptoms.
Post-Traumatic Stress Severity and Impairment as Assessed by the UCLA PTSD Reaction Index for DSM-5 (UCLA-RI-5) - Parent Reported | baseline, week 7, week 15
  Total score ranges from 0 to 73, with a higher score indicating worse symptoms.
Functional Impairment as Assessed by the Columbia Impairment Scale-Parent and Child (CIS-P/C) | baseline, week 7, week 15
  Total score ranges from 0 to 65, with a higher score indicating a worse outcome.

SECONDARY OUTCOMES:
Number of participants with a PTSD Diagnosis as Assessed by the Diagnostic Interview for Anxiety, Mood, and Obsessive-compulsive disorder (OCD) and Related Neuropsychiatric Disorders Child and Adolescent Version (DIAMOND-KID) Clinical Interview | baseline, week 7, week 15
  A PTSD diagnosis using the DIAMOND-KID Clinical Interview is indicated by answering "yes" to the presence of 4 types of PTSD symptoms.
Anxiety as Assessed by the Revised Child Anxiety and Depression Scale (RCADS-C/P) - Anxiety Subscore | baseline, week 15
  Total score ranges from 0 to 111, with a higher score indicating greater symptom severity.
Depression as Assessed by the Revised Child Anxiety and Depression Scale (RCADS-C/P) - Depression Subscore | baseline, week 15
  Total score ranges from 0 to 30, with a higher score indicating greater symptom severity.
Clinical Severity of Trauma Symptoms as Assessed by the Clinical Global Impression-Severity/Improvement (CGI-S/I) Scale | baseline, week 7, week 15
  Total score ranges from 0 (no illness) to 6 (extremely severe), with a higher score indicating a greater severity of trauma symptoms.
Clinical Improvement in Trauma Symptoms as Assessed by the Clinical Global Impression Severity/Improvement (CGI-S/I) Scale | baseline, week 7, week 15
  Total score ranges from 0 to 7, with a higher score indicating a worse outcome. A score of 1, 2 or 3 will be used to indicate treatment response.
Parent Post-Traumatic Stress Syndrome (PTSS) as Assessed by the PTSD Checklist for DSM-5 (PCL-5) | baseline, week 15
  Total score ranges from 0 to 80, with a higher score indicating a worse outcome.
Parent Depression as Assessed by the Patient Health Questionnaire-9 (PHQ-9) | baseline, week 15
  Total score ranges from 0 to 27, with a higher score indicating a worse outcome.
Parent Anxiety as Assessed by the General Anxiety Disorder-7 (GAD-7) Scale | baseline, week 15
  Total score ranges from 0 to 21, with a higher score indicating a worse outcome.
Parent Stress as Assessed by the Perceived Stress Scale (PSS) | baseline, week 15
  Scores range from 18 to 90, with a higher score indicating higher parenting stress.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie K Taylor, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No